CLINICAL TRIAL: NCT00685503
Title: Pilot Study of Intravitreal Injection of Ranibizumab for Macular Telangiectasia With Neovascularization (MACTEL 1)
Brief Title: Ranibizumab Injections to Treat Macular Telangiectasia With New Blood Vessel Growth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080146; 08-EI-0146
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-12

CONDITIONS: Neovascularization
Keywords: Macular Telangiectasia; Vascular Endothelial Growth Factor; Ranibizumab; Neovascularization
MeSH Terms: conditions — Neovascularization, Pathologic | interventions — Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
This study will examine whether the drug ranibizumab (Lucentis) can help prevent vision loss in people with macular telangiectasia, a condition in which new blood vessels grow in the retina at the back of the eye and can leak. Such changes in blood vessels are seen in other diseases associated with changes in a body chemical called vascular endothelial growth factor (VEGF). Ranibizumab is an anti-VEGF drug that is effective in treating another eye disease, age-related macular degeneration, with similar changes in eye blood vessels.

People 18 years of age and older with macular telangiectasia in both eyes and new blood vessel growth in at least one eye may be eligible for this study. They must have vision better than 20/400 in the study eye.

Participants undergo the following procedures:

* Ranibizumab injections in the study eye at least four times over 12 weeks. Depending on the response to treatment and the side effects, additional injections may be given every 4 weeks for up to 1 year. The eye is numbed before the injection and the eye area is cleaned with an antiseptic. Antibiotic drops are used for 3 days following the injection to prevent infection.
* Evaluations before starting treatment, at the time of each injection, and 8 weeks after the last treatment:

  * History and physical examination.
  * Eye examination with dilation, microperimetry and photography: The eye examination measures visual acuity, eye pressure and eye movements. For the microperimetry test, subjects sit in front of a computer screen and press a button when they see a light on the screen. Measurements and photographs of the retina are also taken.
  * Fluorescein and indocyanine green angiography to examine the blood vessels in the eye: A dye called fluorescein or indocyanine green is injected into a vein in the arm. The dye travels through the veins to the blood vessels in the eyes. A camera takes pictures of the dye as it flows through the blood vessels.
  * Pregnancy test: Women who are able to become pregnant have a urine pregnancy test before each ranibizumab injection.

DETAILED DESCRIPTION:
Retinal telangiectasis is a group of rare, idiopathic retinal vascular anomalies affecting the retinal capillaries in which irregular capillary dilation and incompetence occur in the macula. This is group 2 in the Gass classification of idiopathic juxtafoveal telangiectasia in which fluorescein angiography showed leakage with capillary dilation. These patients typically are diagnosed in their fifth or sixth decade of life. Both sexes may be affected. Minimal exudation, superficial retinal crystalline deposits, and right-angle venules characterize this disorder. As the disease progresses, intraretinal pigment plaques and intraretinal and eventually subretinal/choroidal neovascularization develop. The pathogenesis of the disease is unknown. Because of the leakage of the retinal vessels and also the finding of neovascularization, it is possible that vascular endothelial growth factor (VEGF) may be implicated in this disease.

The purpose of this study is to evaluate the possible role of ranibizumab for the treatment of eight participants with macular telangiectasia with hyperfluorescence on fluorescein angiography, with vision better than 20/400, with neovascularization. The primary outcome of this study will be the proportion of participants that lose 15 letters or more in ETDRS BCVA at 12 months compared with baseline. The secondary outcomes measured at one year will include the proportion of participants who lose 10 letters or more, the change in central retinal thickness, the mean change in ETDRS BCVA, the extent of fluorescein leakage, the change in fundus autofluorescence change in size of neovascular membrane, and the change in central retinal sensitivity. This is a pilot study designed to evaluate the feasibility and potential efficacy of treating patients with macular telangiectasia in a larger, phase III study within the organization of the MAC TEL Research Group, sponsored by the Lowy Foundation. Currently, the research group is enrolling 200 patients affected with this condition for a natural history study in 22 international clinical centers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant must understand and sign the informed consent.
* Participant must be at least 18 years of age.
* Participant must have macular telangiectasia in both eyes.
* Participant must have neovascularization in the study eye.
* Participant must have vision loss of better than 20/400 in the study eye.
* Participant must have clear ocular media and adequate pupillary dilation to permit good quality stereoscopic fundus photography.
* All women of childbearing potential must have a negative urine pregnancy test at baseline, and be willing to undergo testing immediately prior to each injection and monthly for at least 2 months following the last dose of ranibizumab.
* Safety and toxicity of ranibizumab have not yet been investigated in children. Further, it is unlikely that younger participants will be able to comply with all examinations and intravitreal injections. Therefore, participants below the age of 18 will be excluded from participation in the study. This ocular condition is not commonly found in participants below the age of 18.

EXCLUSION CRITERIA:

* History (within past five years) of a myocardial infarction or cerebrovascular accident or evidence of severe cardiac disease (apparent in electrocardiogram abnormalities, clinical history of unstable angina, acute coronary syndrome, myocardial infarction, revascularization procedure within six months prior to baseline, atrial or ventricular tachyarrythmias requiring ongoing treatment).
* History of stroke within 12 months of study entry.
* History within the past 30 days of a chronic ocular or periocular infection (including any history of ocular herpes zoster).
* Current acute ocular or periocular infection.
* Any major surgical procedure within one month of study entry.
* Known serious allergies to fluorescein dye AND either indocyanine green dye iodine, or shellfish. Indocyanine green dye is contraindicated in patients with iodine and shellfish allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-05-21; Primary Completion 2011-04-12 (Actual); Study Completion 2011-04-12 (Actual)

PRIMARY OUTCOMES:
Effect of intravitreal ranibizumab treatment on visual acuity.

SECONDARY OUTCOMES:
ETDRS BCVA, area of retinal leakage, retinal thickness, area of hypofluoresence, central retinal sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Amin R, Puklin JE, Frank RN. Growth factor localization in choroidal neovascular membranes of age-related macular degeneration. Invest Ophthalmol Vis Sci. 1994 Jul;35(8):3178-88. PMID 7519180
- [Background] Boulton M, Foreman D, Williams G, McLeod D. VEGF localisation in diabetic retinopathy. Br J Ophthalmol. 1998 May;82(5):561-8. doi: 10.1136/bjo.82.5.561. PMID 9713066